CLINICAL TRIAL: NCT03915860
Title: A Multi-Center Study to Evaluate Subject Reported Outcomes With Use of Trifarotene 50 μg/g Cream in the Treatment of Moderate Facial and Truncal Acne Vulgaris
Brief Title: Participant Reported Outcomes With Use of Trifarotene 50 μg/g Cream in the Treatment of Moderate Facial and Truncal Acne Vulgaris
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RD.06.SPR.118295
Record Dates: First submitted 2019-04-12; First posted 2019-04-16 (Actual); Results first posted 2021-12-15 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2019-04

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — trifarotene

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Trifarotene (Experimental): Participants applied Trifarotene 50 μg/g topically once daily in the evening for 24 weeks.
  Interventions: Drug: Trifarotene

INTERVENTIONS:
Drug: Trifarotene — Topical Cream

SUMMARY:
Participant Reported Outcomes with use of Trifarotene 50 μg/g Cream in participants with Moderate Facial and Truncal Acne Vulgaris

DETAILED DESCRIPTION:
There was no formal hypothesis to be tested. Approximately 50 subjects would be enrolled to evaluate the subject reported outcomes (quality of life and satisfaction survey). The sample size was not based on any formal hypothesis testing.

ELIGIBILITY:
Inclusion Criteria:

* The participant was a male or female, 9 years of age or older, at Screening visit.
* The participant had moderate acne at Screening and Baseline.
* The participant was a female of non childbearing potential.
* The participant was a female of childbearing potential with a negative pregnancy test and who was strictly abstinent or who agreed to use an effective and approved contraceptive method for the duration of the study and at least 1 months after the last study drug application.

Exclusion Criteria:

* The participant had severe forms of acne (e.g., acne conglobate, acne fulminant) or secondary acne form (e.g., chloracne, drug induced acne, etc.).
* The participant had any uncontrolled or serious disease or any medical or surgical condition that may either interfere with the interpretation of the trial results and/or put the participant at significant risk (according to the Investigator's judgment) if the participant took part to the trial.
* The participant had been exposed to excessive ultraviolet (UV) radiation within one month prior to the Baseline visit or the participant was planning intense UV exposure during the study (i.ed, occupational exposure to the sun, sunbathing, tanning salon use, phototherapy, etc.).
* The participant was unwilling to refrain from use of prohibited medication during the Clinical Trial.

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2019-03-27 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2019-12-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Galderma Investigational Site, Fort Smith, Arkansas
  - Galderma Investigational Site, Beverly, Massachusetts
  - Galderma Investigational Site, Portsmouth, New Hampshire
  - Galderma Investigational Site, Philadelphia, Pennsylvania
  - Galderma Investigational Site, Austin, Texas
  - Galderma Investigational Site, Beaumont, Texas
  - Galderma Investigational Site, Irving, Texas
  - Galderma Investigational Site, Pflugerville, Texas
  - Galderma Investigational Site, Richardson, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at United States between 27 March 2019 and 23 December 2019.
Pre-assignment Details: A total of 47 participants were enrolled in the study. Of which, 46 participants were treated.
Period: Overall Study
Arm/Group | Trifarotene
Started | 47
Treated | 46
Completed | 33
Not Completed | 14
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 6
Not completed — Lost to Follow-up | 2
Not completed — Other than specified | 3

BASELINE CHARACTERISTICS:
Population: Analysis was performed on Intent to treat (ITT) population that included all enrolled participants.
Arm/Group | Trifarotene
Number analyzed (Participants) | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.6 (3.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 37
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 42
  More than one race | 0
  Unknown or Not Reported | 0
Dermatology Life Quality Index (DLQI) Score at Baseline [Mean (Standard Deviation); unit: score on a scale] — The DLQI was validated 10-item questionnaire that measured the dermatology-related limitations of functional ability and the frequency, severity, and impact of general inflammatory skin conditions on the quality-of-life (QOL). Total DLQI score was calculated by summing the scores of each question, resulting in a maximum of 30 and minimum of 0. Responses to each questions were assessed on a scale of 0 to 3, where 0="not at all" & 3="very much". Scores from all 10 questions added up to give total DLQI scores ranged from 0(not at all) to 30(very much),higher scores=more impact on quality of life Population: Here, number analyzed=participants with available data at Baseline.
  score on a scale
    number analyzed (Participants) | 13
    (all) | 2.8 (3.00)
C-DLQI (Children's Dermatology Life Quality Index) Score at Baseline [Mean (Standard Deviation); unit: score on a scale] — The C-DLQI are validated 10-item questionnaire that measured the dermatology related limitations of functional ability and the frequency, severity, and impact of general inflammatory skin conditions on the quality-of-life (QOL). Questions were scored as follows: No effect (0-1), Small effect (2-6), Moderate effect (7-12), Very large effect (13-18), Extremely large effect (19-30). The total C-DLQI score was calculated by summing the scores of each question, resulting in a maximum of 30 (Extremely large effect) and a minimum of 0 (No effect). A lower score on the C-DLQI indicates increased QOL. Population: Here, number analyzed=participants with available data at Baseline.
  score on a scale
    number analyzed (Participants) | 33
    (all) | 3.2 (4.17)
Comprehensive Quality of Life (QOL) Measure for Facial and Truncal Acne at Baseline [Mean (Standard Deviation); unit: score on a scale] — The CompAQ questionnaire is a comprehensive measure of facial and truncal acne's impact on health-related QOL. The 20 questions consisted of 5 domains that assessed a variety of psychosocial and physical impacts of acne: Psychological/Emotional, Social (Judgement from Others), Social Interactions, Treatment Concerns, Physical Symptoms. Each question is assessed with a numeric score between 0 (Never) and 8 (All the time) with a total possible score range of 0 (No effect) -160 (greater adverse impact). The higher the score, the more quality of life is impaired. Population: Here, number analyzed=participants with available data at Baseline
  score on a scale
    number analyzed (Participants) | 19
    (all) | 37.8 (17.69)
EuroQoL 5-Dimension (EQ-5D-5L) Index Score at Baseline [Mean (Standard Deviation); unit: score on a scale] — EQ-5D-5L is a 2-part measurement. The first part is comprised of the following 5 participant-reported dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The responses are used to derive the health state index scores using the United States (US) algorithm, with scores ranging from -0.109 (extreme problems) to 1 (no problems). A higher score indicates better health state.
  score on a scale | 0.9416 (0.07334)
EuroQoL 5-Dimension (EQ-5D-5L) VAS Score at Baseline [Mean (Standard Deviation); unit: score on a scale] — The EQ-5D-5L assesses general health-related quality of life. The second portion of the scale is a self-perceived health score assessed using a VAS that ranges from 0 (the worst imaginable health) to 100 (the best imaginable health), with higher scores indicating higher health utility.
  score on a scale | 90.0 (8.99)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) Total Score at Week 12 and 24
Description: The DLQI was validated 10-item questionnaire for participants aged >16 years that measured the dermatology-related limitations of functional ability and the frequency, severity, and impact of general inflammatory skin conditions on the quality-of-life (QOL). The total DLQI score was calculated by summing the scores of each question, resulting in a maximum of 30 and a minimum of 0. Responses to each questions were assessed on a scale of 0 to 3, where 0 is "not at all" and 3 is "very much". Scores from all 10 questions added up to give total DLQI scores ranged from 0 (not at all) to 30 (very much), higher scores indicated more impact on quality of life.
Time Frame: Baseline, Week 12 and Week 24
Population: Analysis was performed on ITT population that included all enrolled participants. Here, overall number of participants analyzed=participants with available data at Week 12 and 24.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Trifarotene
Number analyzed (Participants) | 10
score on a scale
  Week 12 | -1.8 (2.97)
  Week 24 | -0.5 (5.85)

2. Primary Outcome: Change From Baseline in C-DLQI (Children's Dermatology Life Quality Index) Score at Week 12 and 24
Description: The C-DLQI are validated 10-item questionnaire for participants aged <=16 that measured the dermatology related limitations of functional ability and the frequency, severity, and impact of general inflammatory skin conditions on the quality-of-life (QOL). Questions were scored as follows: No effect (0-1), Small effect (2-6), Moderate effect (7-12), Very large effect (13-18), Extremely large effect (19-30). The total C-DLQI score was calculated by summing the scores of each question, resulting in a maximum of 30 (Extremely large effect) and a minimum of 0 (No effect). A lower score on the C-DLQI indicates increased QOL.
Time Frame: Baseline, Week 12 and Week 24
Population: Analysis was performed on ITT population. Here, overall number of participants analyzed=participants with available data at Baseline. Number analyzed=participants with available data at specified time-points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Trifarotene
Number analyzed (Participants) | 33
score on a scale
  Week 12: number analyzed (Participants) | 23
  Week 12 | -1.7 (4.28)
  Week 24: number analyzed (Participants) | 29
  Week 24 | -1.2 (5.03)

3. Primary Outcome: Change From Baseline in Comprehensive Quality of Life (QOL) Measure for Facial and Truncal Acne (CompAQ) Total Score at Week 12, 24
Description: The CompAQ questionnaire is a comprehensive measure of facial and truncal acne's impact on health-related QOL. The 20 questions consisted of 5 domains that assessed a variety of psychosocial and physical impacts of acne: Psychological/Emotional, Social (Judgement from Others), Social Interactions, Treatment Concerns, Physical Symptoms. Each question is assessed with a numeric score between 0 (Never) and 8 (All the time) with a total possible score range of 0 (No effect) -160 (greater adverse impact). The higher the score, the more quality of life is impaired.
Time Frame: Baseline, Week 12 and Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Trifarotene
Number analyzed (Participants) | 19
score on a scale
  Week 12: number analyzed (Participants) | 14
  Week 12 | -7.4 (17.39)
  Week 24: number analyzed (Participants) | 15
  Week 24 | -0.6 (39.96)

4. Primary Outcome: Number of Participants With Satisfaction Questionnaire - Treatment Area Face at Week 12 and 24/End of Treatment (ET)
Description: Participants Satisfaction Questionnaire included questions: a) How bothered were you by treatment side effects? : Not bothered at all, Bothered somewhat, Bothered, Bothered a great deal b) Satisfied with the time it took for treatment to work: Very satisfied, Satisfied, Somewhat satisfied, Not satisfied c) How satisfied were you with the effectiveness of the treatment? Very satisfied, Satisfied, Somewhat satisfied, Not satisfied d) How do you feel about yourself, since starting your treatment?: Very much better, A lot better, A little better, Worse. e) Overall, are you satisfied with the treatment? : Very satisfied, Satisfied, Somewhat satisfied, Not satisfied. f) Would you consider using this treatment again: Yes, No. g) Did you use the provided moisturizing lotion?: Yes, No.
Time Frame: Week 12 and Week 24/End of Treatment (ET)
Population: Analysis was performed on ITT population. Here, "number analyzed"=participants with available data at specified time-points.
Measure: Count of Participants; unit: Participants
Arm/Group | Trifarotene
Number analyzed (Participants) | 47
Participants
  Week 12: Bothered By Treatment Side Effects: Not bothered at all: number analyzed (Participants) | 34
  Week 12: Bothered By Treatment Side Effects: Not bothered at all | 18
  Week 12: Bothered By Treatment Side Effects: Bothered somewhat: number analyzed (Participants) | 34
  Week 12: Bothered By Treatment Side Effects: Bothered somewhat | 15
  Week 12: Bothered By Treatment Side Effects: Bothered: number analyzed (Participants) | 34
  Week 12: Bothered By Treatment Side Effects: Bothered | 0
  Week 12: Bothered By Treatment Side Effects: Bothered a great deal: number analyzed (Participants) | 34
  Week 12: Bothered By Treatment Side Effects: Bothered a great deal | 1
  Week 12: Satisfied with the time it took for treatment to work: Very satisfied: number analyzed (Participants) | 34
  Week 12: Satisfied with the time it took for treatment to work: Very satisfied | 8
  Week 12: Satisfied with the time it took for treatment to work: satisfied: number analyzed (Participants) | 34
  Week 12: Satisfied with the time it took for treatment to work: satisfied | 14
  Week 12: Satisfied with the time it took for treatment to work: Somewhat satisfied: number analyzed (Participants) | 34
  Week 12: Satisfied with the time it took for treatment to work: Somewhat satisfied | 9
  Week 12: Satisfied with the time it took for treatment to work: Not satisfied: number analyzed (Participants) | 34
  Week 12: Satisfied with the time it took for treatment to work: Not satisfied | 3
  Week 12: Satisfied with effectiveness of treatment: Very satisfied: number analyzed (Participants) | 34
  Week 12: Satisfied with effectiveness of treatment: Very satisfied | 5
  Week 12: Satisfied with effectiveness of treatment: satisfied: number analyzed (Participants) | 34
  Week 12: Satisfied with effectiveness of treatment: satisfied | 18
  Week 12: Satisfied with effectiveness of treatment: Somewhat satisfied: number analyzed (Participants) | 34
  Week 12: Satisfied with effectiveness of treatment: Somewhat satisfied | 8
  Week 12: Satisfied with effectiveness of treatment: Not satisfied: number analyzed (Participants) | 34
  Week 12: Satisfied with effectiveness of treatment: Not satisfied | 3
  Week 12: Feel about yourself: Very much better: number analyzed (Participants) | 34
  Week 12: Feel about yourself: Very much better | 5
  Week 12: Feel about yourself: A lot better: number analyzed (Participants) | 34
  Week 12: Feel about yourself: A lot better | 14
  Week 12: Feel about yourself: A little better: number analyzed (Participants) | 34
  Week 12: Feel about yourself: A little better | 13
  Week 12: Feel about yourself: Worse: number analyzed (Participants) | 34
  Week 12: Feel about yourself: Worse | 2
  Week 12: Overall-satisfied with the treatment: Very satisfied: number analyzed (Participants) | 34
  Week 12: Overall-satisfied with the treatment: Very satisfied | 6
  Week 12: Overall-satisfied with the treatment: satisfied: number analyzed (Participants) | 34
  Week 12: Overall-satisfied with the treatment: satisfied | 18
  Week 12: Overall-satisfied with the treatment: Somewhat satisfied: number analyzed (Participants) | 34
  Week 12: Overall-satisfied with the treatment: Somewhat satisfied | 7
  Week 12: Overall-satisfied with the treatment: Not satisfied: number analyzed (Participants) | 34
  Week 12: Overall-satisfied with the treatment: Not satisfied | 3
  Week 12: Would you consider using this treatment again -Yes: number analyzed (Participants) | 34
  Week 12: Would you consider using this treatment again -Yes | 31
  Week 12: Would you consider using this treatment again - No: number analyzed (Participants) | 34
  Week 12: Would you consider using this treatment again - No | 3
  Week 12: Used moisturizing lotion: Yes: number analyzed (Participants) | 34
  Week 12: Used moisturizing lotion: Yes | 32
  Week 12: Used moisturizing lotion: No: number analyzed (Participants) | 34
  Week 12: Used moisturizing lotion: No | 2
  Week 12: Used moisturizing lotion: moisturizer helps to reduce irritation: Yes: number analyzed (Participants) | 32
  Week 12: Used moisturizing lotion: moisturizer helps to reduce irritation: Yes | 23
  Week 12: Used moisturizing lotion: moisturizer helps to reduce irritation: No: number analyzed (Participants) | 32
  Week 12: Used moisturizing lotion: moisturizer helps to reduce irritation: No | 9
  Week 12: Used moisturizing lotion: moisturizer helps you to be adherent to study treatment: Yes: number analyzed (Participants) | 32
  Week 12: Used moisturizing lotion: moisturizer helps you to be adherent to study treatment: Yes | 7
  Week 12: Used moisturizing lotion: moisturizer helps you to be adherent to study treatment: No: number analyzed (Participants) | 32
  Week 12: Used moisturizing lotion: moisturizer helps you to be adherent to study treatment: No | 25
  Week 12: Used moisturizing lotion: moisturizer was pleasant to use: Yes: number analyzed (Participants) | 32
  Week 12: Used moisturizing lotion: moisturizer was pleasant to use: Yes | 15
  Week 12: Used moisturizing lotion: moisturizer was pleasant to use: No: number analyzed (Participants) | 32
  Week 12: Used moisturizing lotion: moisturizer was pleasant to use: No | 17
  Week 12: Used moisturizing lotion: None of the above: Yes: number analyzed (Participants) | 32
  Week 12: Used moisturizing lotion: None of the above: Yes | 2
  Week 12: Used moisturizing lotion: None of the above: No: number analyzed (Participants) | 32
  Week 12: Used moisturizing lotion: None of the above: No | 30
  Week 24/ET: Bothered By Treatment Side Effects: Not bothered at all: number analyzed (Participants) | 39
  Week 24/ET: Bothered By Treatment Side Effects: Not bothered at all | 22
  Week 24/ET: Bothered By Treatment Side Effects: Bothered somewhat: number analyzed (Participants) | 39
  Week 24/ET: Bothered By Treatment Side Effects: Bothered somewhat | 13
  Week 24/ET: Bothered By Treatment Side Effects: Bothered: number analyzed (Participants) | 39
  Week 24/ET: Bothered By Treatment Side Effects: Bothered | 4
  Week 24/ET: Bothered By Treatment Side Effects: Bothered a great deal: number analyzed (Participants) | 39
  Week 24/ET: Bothered By Treatment Side Effects: Bothered a great deal | 0
  Week 24/ET: Satisfied with the time it took for treatment to work: Very satisfied: number analyzed (Participants) | 39
  Week 24/ET: Satisfied with the time it took for treatment to work: Very satisfied | 9
  Week 24/ET: Satisfied with the time it took for treatment to work: satisfied: number analyzed (Participants) | 39
  Week 24/ET: Satisfied with the time it took for treatment to work: satisfied | 20
  Week 24/ET: Satisfied with the time it took for treatment to work: Somewhat satisfied: number analyzed (Participants) | 39
  Week 24/ET: Satisfied with the time it took for treatment to work: Somewhat satisfied | 5
  Week 24/ET: Satisfied with the time it took for treatment to work: Not satisfied: number analyzed (Participants) | 39
  Week 24/ET: Satisfied with the time it took for treatment to work: Not satisfied | 5
  Week 24/ET: Satisfied with effectiveness of treatment: Very satisfied: number analyzed (Participants) | 39
  Week 24/ET: Satisfied with effectiveness of treatment: Very satisfied | 11
  Week 24/ET: Satisfied with effectiveness of treatment: satisfied: number analyzed (Participants) | 39
  Week 24/ET: Satisfied with effectiveness of treatment: satisfied | 15
  Week 24/ET: Satisfied with effectiveness of treatment: Somewhat satisfied: number analyzed (Participants) | 39
  Week 24/ET: Satisfied with effectiveness of treatment: Somewhat satisfied | 8
  Week 24/ET: Satisfied with effectiveness of treatment: Not satisfied: number analyzed (Participants) | 39
  Week 24/ET: Satisfied with effectiveness of treatment: Not satisfied | 5
  Week 24/ET: Feel about yourself: Very much better: number analyzed (Participants) | 39
  Week 24/ET: Feel about yourself: Very much better | 9
  Week 24/ET: Feel about yourself: A lot better: number analyzed (Participants) | 39
  Week 24/ET: Feel about yourself: A lot better | 9
  Week 24/ET: Feel about yourself: A little better: number analyzed (Participants) | 39
  Week 24/ET: Feel about yourself: A little better | 19
  Week 24/ET: Feel about yourself: Worse: number analyzed (Participants) | 39
  Week 24/ET: Feel about yourself: Worse | 2
  Week 24/ET: Overall-satisfied with the treatment: Very satisfied: number analyzed (Participants) | 39
  Week 24/ET: Overall-satisfied with the treatment: Very satisfied | 12
  Week 24/ET: Overall-satisfied with the treatment: satisfied: number analyzed (Participants) | 39
  Week 24/ET: Overall-satisfied with the treatment: satisfied | 12
  Week 24/ET: Overall-satisfied with the treatment: Somewhat satisfied: number analyzed (Participants) | 39
  Week 24/ET: Overall-satisfied with the treatment: Somewhat satisfied | 11
  Week 24/ET: Overall-satisfied with the treatment: Not satisfied: number analyzed (Participants) | 39
  Week 24/ET: Overall-satisfied with the treatment: Not satisfied | 4
  Week 24/ET: Would you consider using this treatment again -Yes: number analyzed (Participants) | 39
  Week 24/ET: Would you consider using this treatment again -Yes | 28
  Week 24/ET: Would you consider using this treatment again - No: number analyzed (Participants) | 39
  Week 24/ET: Would you consider using this treatment again - No | 11
  Week 24/ET: Used moisturizing lotion: Yes: number analyzed (Participants) | 39
  Week 24/ET: Used moisturizing lotion: Yes | 38
  Week 24/ET: Used moisturizing lotion: No: number analyzed (Participants) | 39
  Week 24/ET: Used moisturizing lotion: No | 1
  Week 24/ET: Used moisturizing lotion: moisturizer helps to reduce irritation: Yes: number analyzed (Participants) | 38
  Week 24/ET: Used moisturizing lotion: moisturizer helps to reduce irritation: Yes | 30
  Week 24/ET: Used moisturizing lotion: moisturizer helps to reduce irritation: No: number analyzed (Participants) | 38
  Week 24/ET: Used moisturizing lotion: moisturizer helps to reduce irritation: No | 8
  Week 24/ET: Used moisturizing lotion: moisturizer helps you to be adherent to study treatment: Yes: number analyzed (Participants) | 38
  Week 24/ET: Used moisturizing lotion: moisturizer helps you to be adherent to study treatment: Yes | 7
  Week 24/ET: Used moisturizing lotion: moisturizer helps you to be adherent to study treatment: No: number analyzed (Participants) | 38
  Week 24/ET: Used moisturizing lotion: moisturizer helps you to be adherent to study treatment: No | 31
  Week 24/ET: Used moisturizing lotion: moisturizer was pleasant to use: Yes: number analyzed (Participants) | 38
  Week 24/ET: Used moisturizing lotion: moisturizer was pleasant to use: Yes | 15
  Week 24/ET: Used moisturizing lotion: moisturizer was pleasant to use: No: number analyzed (Participants) | 38
  Week 24/ET: Used moisturizing lotion: moisturizer was pleasant to use: No | 23
  Week 24/ET: Used moisturizing lotion: None of the above: Yes: number analyzed (Participants) | 38
  Week 24/ET: Used moisturizing lotion: None of the above: Yes | 2
  Week 24/ET: Used moisturizing lotion: None of the above: No: number analyzed (Participants) | 38
  Week 24/ET: Used moisturizing lotion: None of the above: No | 36

5. Primary Outcome: Number of Participants With Satisfaction Questionnaire - Treatment Area Trunk at Week 12 and 24/ End of Treatment (ET)
Description: as for outcome 4
Time Frame: Week 12 and Week 24/ET
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Trifarotene
Number analyzed (Participants) | 47
Participants
  Week 12: Bothered By Treatment Side Effects: Not bothered at all: number analyzed (Participants) | 34
  Week 12: Bothered By Treatment Side Effects: Not bothered at all | 23
  Week 12: Bothered By Treatment Side Effects: Bothered somewhat: number analyzed (Participants) | 34
  Week 12: Bothered By Treatment Side Effects: Bothered somewhat | 9
  Week 12: Bothered By Treatment Side Effects: Bothered: number analyzed (Participants) | 34
  Week 12: Bothered By Treatment Side Effects: Bothered | 2
  Week 12: Bothered By Treatment Side Effects: Bothered a great deal: number analyzed (Participants) | 34
  Week 12: Bothered By Treatment Side Effects: Bothered a great deal | 0
  Week 12: Satisfied with the time it took for treatment to work: Very satisfied: number analyzed (Participants) | 34
  Week 12: Satisfied with the time it took for treatment to work: Very satisfied | 8
  Week 12: Satisfied with the time it took for treatment to work: satisfied: number analyzed (Participants) | 34
  Week 12: Satisfied with the time it took for treatment to work: satisfied | 16
  Week 12: Satisfied with the time it took for treatment to work: Somewhat satisfied: number analyzed (Participants) | 34
  Week 12: Satisfied with the time it took for treatment to work: Somewhat satisfied | 8
  Week 12: Satisfied with the time it took for treatment to work: Not satisfied: number analyzed (Participants) | 34
  Week 12: Satisfied with the time it took for treatment to work: Not satisfied | 2
  Week 12: Satisfied with effectiveness of treatment: Very satisfied: number analyzed (Participants) | 34
  Week 12: Satisfied with effectiveness of treatment: Very satisfied | 5
  Week 12: Satisfied with effectiveness of treatment: satisfied: number analyzed (Participants) | 34
  Week 12: Satisfied with effectiveness of treatment: satisfied | 18
  Week 12: Satisfied with effectiveness of treatment: Somewhat satisfied: number analyzed (Participants) | 34
  Week 12: Satisfied with effectiveness of treatment: Somewhat satisfied | 10
  Week 12: Satisfied with effectiveness of treatment: Not satisfied: number analyzed (Participants) | 34
  Week 12: Satisfied with effectiveness of treatment: Not satisfied | 1
  Week 12: Feel about yourself: Very much better: number analyzed (Participants) | 34
  Week 12: Feel about yourself: Very much better | 6
  Week 12: Feel about yourself: A lot better: number analyzed (Participants) | 34
  Week 12: Feel about yourself: A lot better | 14
  Week 12: Feel about yourself: A little better: number analyzed (Participants) | 34
  Week 12: Feel about yourself: A little better | 14
  Week 12: Feel about yourself: Worse: number analyzed (Participants) | 34
  Week 12: Feel about yourself: Worse | 0
  Week 12: Overall-satisfied with the treatment: Very satisfied: number analyzed (Participants) | 34
  Week 12: Overall-satisfied with the treatment: Very satisfied | 8
  Week 12: Overall-satisfied with the treatment: satisfied: number analyzed (Participants) | 34
  Week 12: Overall-satisfied with the treatment: satisfied | 13
  Week 12: Overall-satisfied with the treatment: Somewhat satisfied: number analyzed (Participants) | 34
  Week 12: Overall-satisfied with the treatment: Somewhat satisfied | 10
  Week 12: Overall-satisfied with the treatment: Not satisfied: number analyzed (Participants) | 34
  Week 12: Overall-satisfied with the treatment: Not satisfied | 3
  Week 12: Would you consider using this treatment again -Yes: number analyzed (Participants) | 34
  Week 12: Would you consider using this treatment again -Yes | 32
  Week 12: Would you consider using this treatment again - No: number analyzed (Participants) | 34
  Week 12: Would you consider using this treatment again - No | 2
  Week 12: Used moisturizing lotion: Yes: number analyzed (Participants) | 34
  Week 12: Used moisturizing lotion: Yes | 33
  Week 12: Used moisturizing lotion: No: number analyzed (Participants) | 34
  Week 12: Used moisturizing lotion: No | 1
  Week 12: Used moisturizing lotion: moisturizer helps to reduce irritation: Yes: number analyzed (Participants) | 33
  Week 12: Used moisturizing lotion: moisturizer helps to reduce irritation: Yes | 23
  Week 12: Used moisturizing lotion: moisturizer helps to reduce irritation: No: number analyzed (Participants) | 33
  Week 12: Used moisturizing lotion: moisturizer helps to reduce irritation: No | 10
  Week 12: Used moisturizing lotion: moisturizer helps you to be adherent to study treatment: Yes: number analyzed (Participants) | 33
  Week 12: Used moisturizing lotion: moisturizer helps you to be adherent to study treatment: Yes | 8
  Week 12: Used moisturizing lotion: moisturizer helps you to be adherent to study treatment: No: number analyzed (Participants) | 33
  Week 12: Used moisturizing lotion: moisturizer helps you to be adherent to study treatment: No | 25
  Week 12: Used moisturizing lotion: moisturizer was pleasant to use: Yes: number analyzed (Participants) | 33
  Week 12: Used moisturizing lotion: moisturizer was pleasant to use: Yes | 14
  Week 12: Used moisturizing lotion: moisturizer was pleasant to use: No: number analyzed (Participants) | 33
  Week 12: Used moisturizing lotion: moisturizer was pleasant to use: No | 19
  Week 12: Used moisturizing lotion: None of the above: Yes: number analyzed (Participants) | 33
  Week 12: Used moisturizing lotion: None of the above: Yes | 3
  Week 12: Used moisturizing lotion: None of the above: No: number analyzed (Participants) | 33
  Week 12: Used moisturizing lotion: None of the above: No | 30
  Week 24/ET: Bothered By Treatment Side Effects: Not bothered at all: number analyzed (Participants) | 39
  Week 24/ET: Bothered By Treatment Side Effects: Not bothered at all | 22
  Week 24/ET: Bothered By Treatment Side Effects: Bothered somewhat: number analyzed (Participants) | 39
  Week 24/ET: Bothered By Treatment Side Effects: Bothered somewhat | 13
  Week 24/ET: Bothered By Treatment Side Effects: Bothered: number analyzed (Participants) | 39
  Week 24/ET: Bothered By Treatment Side Effects: Bothered | 4
  Week 24/ET: Bothered By Treatment Side Effects: Bothered a great deal: number analyzed (Participants) | 39
  Week 24/ET: Bothered By Treatment Side Effects: Bothered a great deal | 0
  Week 24/ET: Satisfied with the time it took for treatment to work: Very satisfied: number analyzed (Participants) | 39
  Week 24/ET: Satisfied with the time it took for treatment to work: Very satisfied | 7
  Week 24/ET: Satisfied with the time it took for treatment to work: satisfied: number analyzed (Participants) | 39
  Week 24/ET: Satisfied with the time it took for treatment to work: satisfied | 22
  Week 24/ET: Satisfied with the time it took for treatment to work: Somewhat satisfied: number analyzed (Participants) | 39
  Week 24/ET: Satisfied with the time it took for treatment to work: Somewhat satisfied | 5
  Week 24/ET: Satisfied with the time it took for treatment to work: Not satisfied: number analyzed (Participants) | 39
  Week 24/ET: Satisfied with the time it took for treatment to work: Not satisfied | 5
  Week 24/ET: Satisfied with effectiveness of treatment: Very satisfied: number analyzed (Participants) | 39
  Week 24/ET: Satisfied with effectiveness of treatment: Very satisfied | 8
  Week 24/ET: Satisfied with effectiveness of treatment: satisfied: number analyzed (Participants) | 39
  Week 24/ET: Satisfied with effectiveness of treatment: satisfied | 19
  Week 24/ET: Satisfied with effectiveness of treatment: Somewhat satisfied: number analyzed (Participants) | 39
  Week 24/ET: Satisfied with effectiveness of treatment: Somewhat satisfied | 7
  Week 24/ET: Satisfied with effectiveness of treatment: Not satisfied: number analyzed (Participants) | 39
  Week 24/ET: Satisfied with effectiveness of treatment: Not satisfied | 5
  Week 24/ET: Feel about yourself: Very much better: number analyzed (Participants) | 39
  Week 24/ET: Feel about yourself: Very much better | 8
  Week 24/ET: Feel about yourself: A lot better: number analyzed (Participants) | 39
  Week 24/ET: Feel about yourself: A lot better | 11
  Week 24/ET: Feel about yourself: A little better: number analyzed (Participants) | 39
  Week 24/ET: Feel about yourself: A little better | 19
  Week 24/ET: Feel about yourself: Worse: number analyzed (Participants) | 39
  Week 24/ET: Feel about yourself: Worse | 1
  Week 24/ET: Overall-satisfied with the treatment: Very satisfied: number analyzed (Participants) | 39
  Week 24/ET: Overall-satisfied with the treatment: Very satisfied | 10
  Week 24/ET: Overall-satisfied with the treatment: satisfied: number analyzed (Participants) | 39
  Week 24/ET: Overall-satisfied with the treatment: satisfied | 17
  Week 24/ET: Overall-satisfied with the treatment: Somewhat satisfied: number analyzed (Participants) | 39
  Week 24/ET: Overall-satisfied with the treatment: Somewhat satisfied | 9
  Week 24/ET: Overall-satisfied with the treatment: Not satisfied: number analyzed (Participants) | 39
  Week 24/ET: Overall-satisfied with the treatment: Not satisfied | 3
  Week 24/ET: Would you consider using this treatment again -Yes: number analyzed (Participants) | 39
  Week 24/ET: Would you consider using this treatment again -Yes | 28
  Week 24/ET: Would you consider using this treatment again - No: number analyzed (Participants) | 39
  Week 24/ET: Would you consider using this treatment again - No | 11
  Week 24/ET: Used moisturizing lotion: Yes: number analyzed (Participants) | 39
  Week 24/ET: Used moisturizing lotion: Yes | 37
  Week 24/ET: Used moisturizing lotion: No: number analyzed (Participants) | 39
  Week 24/ET: Used moisturizing lotion: No | 2
  Week 24/ET: Used moisturizing lotion: moisturizer helps to reduce irritation: Yes: number analyzed (Participants) | 37
  Week 24/ET: Used moisturizing lotion: moisturizer helps to reduce irritation: Yes | 30
  Week 24/ET: Used moisturizing lotion: moisturizer helps to reduce irritation: No: number analyzed (Participants) | 37
  Week 24/ET: Used moisturizing lotion: moisturizer helps to reduce irritation: No | 7
  Week 24/ET: Used moisturizing lotion: moisturizer helps you to be adherent to study treatment: Yes: number analyzed (Participants) | 37
  Week 24/ET: Used moisturizing lotion: moisturizer helps you to be adherent to study treatment: Yes | 8
  Week 24/ET: Used moisturizing lotion: moisturizer helps you to be adherent to study treatment: No: number analyzed (Participants) | 37
  Week 24/ET: Used moisturizing lotion: moisturizer helps you to be adherent to study treatment: No | 29
  Week 24/ET: Used moisturizing lotion: moisturizer was pleasant to use: Yes: number analyzed (Participants) | 37
  Week 24/ET: Used moisturizing lotion: moisturizer was pleasant to use: Yes | 13
  Week 24/ET: Used moisturizing lotion: moisturizer was pleasant to use: No: number analyzed (Participants) | 37
  Week 24/ET: Used moisturizing lotion: moisturizer was pleasant to use: No | 24
  Week 24/ET: Used moisturizing lotion: None of the above: Yes: number analyzed (Participants) | 37
  Week 24/ET: Used moisturizing lotion: None of the above: Yes | 2
  Week 24/ET: Used moisturizing lotion: None of the above: No: number analyzed (Participants) | 37
  Week 24/ET: Used moisturizing lotion: None of the above: No | 35

6. Primary Outcome: Change From Baseline in EQ-5D-5L Index Score at Week 12 and 24
Description: EQ-5D-5L is a 2-part measurement. The first part is comprised of the following 5 participant-reported dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The responses are used to derive the health state index scores using the United States (US) algorithm, with scores ranging from -0.109 (extreme problems) to 1 (no problems). A higher score indicates better health state.
Time Frame: Baseline, Week 12 and Week 24
Population: Analysis was performed on ITT population. Here, number analyzed=participants with available data at specified time-points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Trifarotene
Number analyzed (Participants) | 47
score on a scale
  Week 12: number analyzed (Participants) | 34
  Week 12 | -0.0140 (0.09626)
  Week 24: number analyzed (Participants) | 40
  Week 24 | 0.0135 (0.08394)

7. Primary Outcome: Change From Baseline in EQ-5D-5L VAS at Week 12 and 24
Description: The EQ-5D-5L assesses general health-related quality of life. The second portion of the scale is a self-perceived health score assessed using a VAS that ranges from 0 (the worst imaginable health) to 100 (the best imaginable health), with higher scores indicating higher health utility.
Time Frame: Baseline, Week 12 and Week 24
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Trifarotene
Number analyzed (Participants) | 47
score on a scale
  Week 12: number analyzed (Participants) | 34
  Week 12 | 1.0 (8.96)
  Week 24: number analyzed (Participants) | 40
  Week 24 | 3.7 (7.96)

8. Secondary Outcome: Percentage of Participants Who Achieved an IGA Score of 1 (Almost Clear) or 0 (Clear) and At Least a 2-Grade Improvement From Baseline to Week 12 and Week 24
Description: IGA was an assessment scale used to evaluate facial acne severity. IGA was recorded from components collected on the case report form (CRF) using a 5-point scale where (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe) based on inflammation, pustules and papulation/infiltration. Success Rate was defined as the percentage of participants who achieved an IGA score of 1 (Almost Clear) or 0 (Clear) and at least a 2-grade improvement from Baseline to Week 12 and Week 24.
Time Frame: Baseline, Week 12 and Week 24
Population: Analysis was performed on Intent-to-treat (ITT) population that included all enrolled participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trifarotene
Number analyzed (Participants) | 47
percentage of participants
  Week 12 | 6.4 [1.3 to 17.5]
  Week 24 | 19.1 [9.1 to 33.3]

9. Secondary Outcome: Percentage of Participants With Physician's Global Assessment of Truncal Acne Success Rate at Week 12 and 24
Description: The Physician's Global Assessment (PGA) was an instrument to evaluate the truncal acne severity in the shoulders, upper back and upper anterior chest areas. PGA was recorded from components collected on the CRF using a 5-point scale where (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe) based on inflammation, pustules and papulation/infiltration. Success Rate was defined as the percentage of participants who achieved an PGA score of 1 (Almost Clear) or 0 (Clear) and at least a 2-grade improvement from Baseline to Week 12 and Week 24. All missing values were imputed by LOCF.
Time Frame: Week 12 and 24
Population: Analysis was performed on Intent-to-treat on the Trunk (ITTT) population that included any participants who were enrolled with moderate truncal acne at the Baseline visit.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trifarotene
Number analyzed (Participants) | 47
percentage of participants
  Week 12 | 14.9 [6.2 to 28.3]
  Week 24 | 6.4 [1.3 to 17.5]

10. Secondary Outcome: Percent Change From Baseline in Facial Inflammatory and Non-inflammatory Lesion Count at Week 12 and 24
Description: Percent change from Baseline was calculated as the values at Week 12 (and 24) minus the value at Baseline divided by Baseline value * 100. All missing values were imputed by LOCF.
Time Frame: Baseline, Week 12 and 24
Population: Analysis was performed on ITT population.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Trifarotene
Number analyzed (Participants) | 47
percent change
  Inflammatory Lesion: Week 12 | -35.81 (41.124)
  Inflammatory Lesion: Week 24 | -38.59 (42.643)
  Non-Inflammatory Lesion: Week 12 | -23.17 (45.506)
  Non-Inflammatory Lesion: Week 24 | -35.16 (46.946)

11. Secondary Outcome: Percent Change From Baseline in Trunk Inflammatory and Non-inflammatory Lesion Count at Week 12 and 24
Description: as for outcome 10
Time Frame: Baseline, Week 12 and Week 24
Population: Analysis was performed on ITT population.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Trifarotene
Number analyzed (Participants) | 47
percent change
  Inflammatory Lesion: Week 12 | -39.97 (32.564)
  Inflammatory Lesion: Week 24 | -41.36 (39.131)
  Non-Inflammatory Lesion: Week 12 | -35.24 (39.337)
  Non-Inflammatory Lesion: Week 24 | -44.20 (37.650)

ADVERSE EVENTS:
Time Frame: From start of the study drug administration up to end of the study (Week 24).
Description: Analysis was performed on Safety Population that included any enrolled participants who applied/were administered the study drug at least once.
Arm/Group | Trifarotene
All-Cause Mortality (participants affected / at risk) | 0/46
Serious Adverse Events (participants affected / at risk) | 0/46
Other Adverse Events (participants affected / at risk) | 9/46
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trifarotene (N=46)
Application site pain (General disorders) | 5 (10)
Application site dermatitis (General disorders) | 3 (3)
Sunburn (Injury, poisoning and procedural complications) | 3 (3)

LIMITATIONS AND CAVEATS:
Small sample size (no formal sample size calculation).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2019-06-04): https://cdn.clinicaltrials.gov/large-docs/60/NCT03915860/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-04): https://cdn.clinicaltrials.gov/large-docs/60/NCT03915860/SAP_001.pdf